CLINICAL TRIAL: NCT04824573
Title: The Effect of Manual Therapy Approaches and Inspiratory Muscle Training on Respiratory Parameters in Healthy Individuals With Hyperkyphosis
Brief Title: Effects of Manual Therapy and Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Şeyda YILDIZ, Research Assistant, Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1700897
Record Dates: First submitted 2021-03-06; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Function
Keywords: inspiration; kyphosis; manual therapy; posture; respiratory muscles
MeSH Terms: conditions — Respiratory Aspiration; Kyphosis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into Inspiratory Muscle Training (IMT) and Manual Therapy groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Experimental): The program of the IMT group (n=16) consists of individual sessions of approximately 20 minutes and the Powerbreathe device (IMT Technologies Ltd., Birmingham) was used for training.
  Interventions: Device: Inspiratory Muscle Training
- Manual Therapy (Experimental): In the manual therapy group (n=19), in addition to the approaches applied to the individuals in the IMT group, a total of eight sessions of manual therapy (manipulation, joint mobilization, and soft tissue mobilization) approaches, two days a week for four weeks and at least two days between sessions, were applied by an experienced physiotherapist in manual therapy. Manual therapy applications; included techniques targeting the cervical and thoracic regions. Techniques for the thoracic region; while it consists of manual diaphragm release, thoracic mobilization and High Velocity Low Amplitude (HVLA) thrust manipulation; the techniques applied to the cervical region consisted of soft tissue and joint mobilization.
  Interventions: Device: Inspiratory Muscle Training; Other: Manual Therapy

INTERVENTIONS:
Device: Inspiratory Muscle Training — Inspiratory Muscle Training (IMT) was performed with Powerbreathe Classic-Light Resistance device. To determine the intensity of the training, MIP values were measured with the help of the respiratory pressure meter-RP Check (MD Diagnostics Ltd. RP Check MIP & MEP) device before each training. The pressure corresponding to 50 percent of the MIP value in the Powerbreathe device was determined as training workload. It was applied two days a week for four weeks, with five-set and five repetitions, for 20 minutes with 30 seconds rest in between. This inspiratory muscle training program has previously been used by several studies to improve respiratory muscle strength.
Other: Manual Therapy — In the manual diaphragm release technique; While the participant was breathing in, the physiotherapist raised his hand slowly to accompany the rising movement of the ribs and deepened the contact during exhalation. The maneuver was performed in two sets of 10 deep breaths.
  In thoracic mobilization application; The physiotherapist, standing behind the participant, wrapped the crossed arms from his right upper arm with his left hand and performed stretching, extension, lateral flexion, and thoracic rotation with his right hand.
  In HVLA thoracic manipulation; the physiotherapist, with the support hand on the participant's elbows, applied HVLA thrust in the posterior-anterior and inferior-superior directions with the help of his body while the manipulating hand was on the transverse processes.
  For cervical joint mobilization; the physiotherapist was applied using the right hand in flexion, extension, right-left rotation, and lateral flexion directions.
  Arms: Manual Therapy

SUMMARY:
The effectiveness of inspiratory muscle training (IMT) and manual therapy approaches added to the IMT program in healthy individuals with hyperkyphosis is uncertain. This study was aimed to determine the effects of manual therapy techniques added to IMT and IMT on pulmonary functions (FVC, FEV1, FEV1 / FVC, and PEF), forward head posture, and hyperkyphosis in healthy individuals with hyperkyphosis. Thirty-five individuals voluntarily participate to study were randomly divided into IMT and manual therapy groups. While all participants received twenty minutes of IMT twice a week for four weeks, manual therapy techniques were applied to the manual therapy group in addition to IMT. Pulmonary functions, forward head posture, and hyperkyphosis were evaluated before and after the treatments with spirometry device; cervical range of joint range of motion measuring device (CROM Deluxe), C0-wall (OWD), and C7-wall distance measurement respectively. Statistical Package for Social Sciences (SPSS 25.0) will be used to analyze the data in the research.

DETAILED DESCRIPTION:
Hyperkyphosis, which is defined as a thoracic curvature higher than normal limits, is among the reasons that decrease chest wall mobility and lung function. In modern society, kyphosis in the thoracic vertebra increases with the increase in sitting time of people. It has been identified in studies that an increase in thoracic kyphosis and a decrease in the mobility of the thoracic region of the spine are associated with a decrease in respiratory functions such as Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1).

Manual therapy approaches consisting of different techniques (manipulation, joint mobilization and soft tissue mobilization) can be an effective approach to improve pulmonary function by increasing chest wall mobility. Manual therapy techniques applied to the thoracic region have been shown to cause a significant reduction in thoracic kyphosis. In a study, it has been shown that thoracic joint mobilization is effective in increasing FVC, FEV1 and Peak Expiratory Flow (PEF) in people with hyperkhyphosis and chronic neck pain. In addition, identified studies shows that manual therapy approaches applied to improve respiratory functions should include both the thoracic and cervical regions due to the relationship between cervical and thoracic spine movements.

Inspiratory Muscle Training (IMT) leads among the approaches used in the current literature to increase respiratory functions. There is important evidence that this technique which aims to increase the strength or endurance of the diaphragm and respiratory assist muscles activated during inspiration, improves respiratory function in the patient and healthy population. In the literature, there are studies examining the effects of IMT and manual therapy approaches on respiratory functions in individuals with chronic obstructive pulmonary disease (COPD), asthma and smokers. In a study conducted on smokers, the effects of manual therapy added to the IMT program on maximum inspiratory pressure (MIP) and other respiratory parameters were examined and a significant increase in MIP was observed, but a significant increase in other respiratory parameters not observed. In another study, it was stated that the addition of manual therapy and therapeutic exercise protocol to IMT in asthmatic individuals was more effective than IMT in improving forward head posture and kyphotic posture.

Although the studies on the effects of using IMT and manual therapy techniques together in healthy individuals on respiratory functions are very limited in the literature, more acute effects were investigated in these studies. In this context, the aim of our study is to evaluate the cervical and thoracic region manual therapy approaches added to IMT and IMT program in healthy individuals with hyperkyphosis; It is the determination of the effects on respiratory function values such as FVC, FEV1, tiffeneau index (FEV1 / FVC) and PEF, forward head posture and hyperkyphosis.

ELIGIBILITY:
Inclusion Criteria:

* individuals who were actively enrolled in Istanbul Esenyurt University
* those who agree to volunteer
* those between the ages of 18-24
* non-smokers
* those with hyperkyphosis
* those with a low physical activity level

Exclusion Criteria:

* those who have moderate or high levels of physical activity
* smokers
* those with a history of traumatic deformity in the thoracic spine
* those who have taken oral corticosteroids or antibiotics within one month
* those diagnosed with scoliosis of 20 ° and above
* those who have had cervical trauma, cervical spine surgery
* those with respiratory system disorders (asthma, etc.)
* those with the meningeal tumor, vertebral tumor, spinal cord tumor, and similar tumors
* individuals with systemic ailments(heart disease, diabetes, hypertension, etc.)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Occiput Wall Distance (OWD) | Change between baseline and 4 weeks
  Participants were asked to touch their occiput against the wall with their back and heels resting touch the wall and head facing forward.
  The presence of hyperkyphosis was considered positive if the wall could not be touched with the occiput.
Forward Head Posture (cm) | Change between baseline and 4 weeks
  The participants were sitting upright on the chair with their arms free at their sides and their feet touching the floor.
  Participants were initially instructed to "sit in a comfortable, natural posture defined as the typical posture you take during your daily activities and do not move your head".
  The head forward arm was attached to the CROM mainframe and the lower end of the control arm (vertebra locator) was held by the investigator on the C7 spinous process.
  The vertebra locator was placed at a 90 ° angle with the forward arm of the CROM with the help of a bubble indicating that the instrument was straight.
  The value on the head forward arm measures the distance in centimeters(cm) between the participant's bridge of nose and C7.
  This measurement was repeated three times in total and the average values were recorded in centimeters(cm)
FEV1 (lt): Forced Expiratory Volume in 1 second | Change between baseline and 4 weeks
  MicroQuark (COSMED, Albano Laziale, Italy) USB spirometer was used for the measurement of FEV1 (lt) measurements.
C7-wall distance measurement (cm) | Change between baseline and 4 weeks
  It is a valid and reliable method of testing performed by measuring the perpendicular distance from the C7 spinous process to the wall.
  The measurement was repeated three times in a row with a short rest period and the mean values were recorded in centimeters (cm)
FVC(lt): Forced vital capacity | Change between baseline and 4 weeks
  MicroQuark (COSMED, Albano Laziale, Italy) USB spirometer was used for the measurement of FVC (lt) measurements.
FEV1/FVC(%): Tiffenea index | Change between baseline and 4 weeks
  MicroQuark (COSMED, Albano Laziale, Italy) USB spirometer was used for the measurement of FVC (lt) measurements.
PEF(lt/sn): Peak expiratory flow | Change between baseline and 4 weeks
  MicroQuark (COSMED, Albano Laziale, Italy) USB spirometer was used for the measurement of FVC (lt) measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla ATAŞ BALCI, Assist Prof., Study Director — Bahçeşehir University; Seçil ÖZKURT, Assist Prof., Study Director — Istanbul Arel University
Locations (1):
- Istanbul Esenyurt University, Istanbul, Esenyurt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwangbo PN, Hwangbo G, Park J, Lee S. The Effect of Thoracic Joint Mobilization and Self-stretching Exercise on Pulmonary Functions of Patients with Chronic Neck Pain. J Phys Ther Sci. 2014 Nov;26(11):1783-6. doi: 10.1589/jpts.26.1783. Epub 2014 Nov 13. PMID 25435700
- [Background] Yaman O, Dalbayrak S. Kyphosis and review of the literature. Turk Neurosurg. 2014;24(4):455-65. doi: 10.5137/1019-5149.JTN.8940-13.0. PMID 25050667
- [Background] Lorbergs AL, O'Connor GT, Zhou Y, Travison TG, Kiel DP, Cupples LA, Rosen H, Samelson EJ. Severity of Kyphosis and Decline in Lung Function: The Framingham Study. J Gerontol A Biol Sci Med Sci. 2017 May 1;72(5):689-694. doi: 10.1093/gerona/glw124. PMID 27341855
- [Background] Wall BA, Peiffer JJ, Losco B, Hebert JJ. The effect of manual therapy on pulmonary function in healthy adults. Sci Rep. 2016 Sep 12;6:33244. doi: 10.1038/srep33244. PMID 27616562
- [Background] Lopez-de-Uralde-Villanueva I, Candelas-Fernandez P, de-Diego-Cano B, Minguez-Calzada O, Del Corral T. The effectiveness of combining inspiratory muscle training with manual therapy and a therapeutic exercise program on maximum inspiratory pressure in adults with asthma: a randomized clinical trial. Clin Rehabil. 2018 Jun;32(6):752-765. doi: 10.1177/0269215517751587. Epub 2018 Jan 10. PMID 29318917
- [Background] Engel RM, Vemulpad S. The effect of combining manual therapy with exercise on the respiratory function of normal individuals: a randomized control trial. J Manipulative Physiol Ther. 2007 Sep;30(7):509-13. doi: 10.1016/j.jmpt.2007.07.006. PMID 17870419
- [Background] Jang SH, Bang HS. Effect of thoracic and cervical joint mobilization on pulmonary function in stroke patients. J Phys Ther Sci. 2016 Jan;28(1):257-60. doi: 10.1589/jpts.28.257. Epub 2016 Jan 30. PMID 26957769
- [Background] Yilmaz Yelvar GD, Cirak Y, Demir YP, Dalkilinc M, Bozkurt B. Immediate effect of manual therapy on respiratory functions and inspiratory muscle strength in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2016 Jun 20;11:1353-7. doi: 10.2147/COPD.S107408. eCollection 2016. PMID 27382271
- [Background] Kim SY, Kim NS, Kim LJ. Effects of cervical sustained natural apophyseal glide on forward head posture and respiratory function. J Phys Ther Sci. 2015 Jun;27(6):1851-4. doi: 10.1589/jpts.27.1851. Epub 2015 Jun 30. PMID 26180334
- [Background] Shei RJ, Paris HL, Wilhite DP, Chapman RF, Mickleborough TD. The role of inspiratory muscle training in the management of asthma and exercise-induced bronchoconstriction. Phys Sportsmed. 2016 Nov;44(4):327-334. doi: 10.1080/00913847.2016.1176546. Epub 2016 Apr 26. PMID 27094568
- [Background] Bostanci O, Mayda H, Yilmaz C, Kabadayi M, Yilmaz AK, Ozdal M. Inspiratory muscle training improves pulmonary functions and respiratory muscle strength in healthy male smokers. Respir Physiol Neurobiol. 2019 Jun;264:28-32. doi: 10.1016/j.resp.2019.04.001. Epub 2019 Apr 3. PMID 30953791
- [Background] Lorenzo S, Nicotra CM, Mentreddy AR, Padia HJ, Stewart DO, Hussein MO, Quinn TA. Assessment of Pulmonary Function After Osteopathic Manipulative Treatment vs Standard Pulmonary Rehabilitation in a Healthy Population. J Am Osteopath Assoc. 2019 Feb 11. doi: 10.7556/jaoa.2019.026. Online ahead of print. PMID 30741314
- [Background] Goosey-Tolfrey V, Foden E, Perret C, Degens H. Effects of inspiratory muscle training on respiratory function and repetitive sprint performance in wheelchair basketball players. Br J Sports Med. 2010 Jul;44(9):665-8. doi: 10.1136/bjsm.2008.049486. Epub 2008 Jul 4. PMID 18603575
- [Background] Cahalin LP, Arena R. Novel methods of inspiratory muscle training via the Test of Incremental Respiratory Endurance (TIRE). Exerc Sport Sci Rev. 2015 Apr;43(2):84-92. doi: 10.1249/JES.0000000000000042. PMID 25607279
- [Background] Balbas-Alvarez L, Candelas-Fernandez P, Del Corral T, La Touche R, Lopez-de-Uralde-Villanueva I. Effect of Manual Therapy, Motor Control Exercise, and Inspiratory Muscle Training on Maximum Inspiratory Pressure and Postural Measures in Moderate Smokers: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2018 Jun;41(5):372-382. doi: 10.1016/j.jmpt.2017.11.004. Epub 2018 Jul 9. PMID 30001903
- [Background] Amatachaya P, Wongsa S, Sooknuan T, Thaweewannakij T, Laophosri M, Manimanakorn N, Amatachaya S. Validity and reliability of a thoracic kyphotic assessment tool measuring distance of the seventh cervical vertebra from the wall. Hong Kong Physiother J. 2016 Jul 13;35:30-36. doi: 10.1016/j.hkpj.2016.05.001. eCollection 2016 Dec. PMID 30931031
- [Background] Garrett TR, Youdas JW, Madson TJ. Reliability of measuring forward head posture in a clinical setting. J Orthop Sports Phys Ther. 1993 Mar;17(3):155-60. doi: 10.2519/jospt.1993.17.3.155. PMID 8472080
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Sonetti DA, Wetter TJ, Pegelow DF, Dempsey JA. Effects of respiratory muscle training versus placebo on endurance exercise performance. Respir Physiol. 2001 Sep;127(2-3):185-99. doi: 10.1016/s0034-5687(01)00250-x. PMID 11504589
- [Background] Volianitis S, McConnell AK, Koutedakis Y, McNaughton L, Backx K, Jones DA. Inspiratory muscle training improves rowing performance. Med Sci Sports Exerc. 2001 May;33(5):803-9. doi: 10.1097/00005768-200105000-00020. PMID 11323552
- [Background] Romer LM, McConnell AK, Jones DA. Effects of inspiratory muscle training on time-trial performance in trained cyclists. J Sports Sci. 2002 Jul;20(7):547-62. doi: 10.1080/026404102760000053. PMID 12166881